CLINICAL TRIAL: NCT00046085
Title: Online Family Support and Education for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH062135 (NIH); R21MH062135 (NIH); DSIR AT-SP
Record Dates: First submitted 2002-09-19; First posted 2002-09-23 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Family; Psychoeducation; Internet
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient customary care (Active Comparator): 12 months of patient customary care
  Interventions: Behavioral: Customary care
- Online family education (Experimental): 12 months of patient customary care and relative access to online education and support program
  Interventions: Behavioral: Online Family Education; Behavioral: Customary care

INTERVENTIONS:
Behavioral: Online Family Education — Families were provided with private, secure access to the website, which features family-to-family chat capabilities, video lectures on the management of schizophrenia, written materials on important issues in schizophrenia management, professionally facilitated online discussions of the material, and additional resource links.
  Arms: Online family education
Behavioral: Customary care — Participants received care as usual.

SUMMARY:
This study evaluated the benefits of providing relatives of patients diagnosed with schizophrenia the opportunity to interact with each other using the Internet. It was hypothesized that patients whose relatives had access to the internet intervention would have reduced symptoms and greater community tenure, compared to their counterparts who did not have relative access to the internet education and support program. We also collected information on how frequently the relatives used the website and how well they liked its features.

DETAILED DESCRIPTION:
Although psychoeducational programs for schizophrenia can reduce patient relapse rates and reduce family distress, participation rates are often low. This study evaluated an online model to provide the families of schizophrenia patients with knowledge of illness management to reduce family burden and increase perceived social support.

Relatives of patients with schizophrenia who received 12 months of customary care with access to the educational website for the first year were compared to matched group of relatives of individuals diagnosed with schizophrenia who were receiving customary care and who consented to participate in a family education program. In the education condition, relatives were provided with private, secure access to the website, which features family-to-family chat capabilities, video lectures on the management of schizophrenia, written materials on important issues in schizophrenia management, professionally facilitated online discussions of the material, and additional resource links.

Relatives were assessed using 90-minute interviews at the beginning of the project and every 6 months for 12 months. The interviews were used to assess the family member's perception of the patient's symptoms, his or her knowledge of the illness, the illness's impact on the family member, and his or her perception of the website intervention.

Patients with schizophrenia or schizoaffective disorder were also asked to complete interviews and assessments at the beginning of the project and every 6 months for 12 months. The assessments include questions about symptoms, medication compliance and side effects, hospitalizations, and social functioning.

The major hypotheses were that relative participation in the online program would be associated with lower symptoms rates and hospitalizations in the patients.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Diagnostic and Statistical Manual (DSM-IV) research diagnosis of schizophrenia or schizoaffective disorder
* Stable antipsychotic medication regimen for at least 1 month
* Willing to participate in in-person assessments

Inclusion Criteria for Relatives:

* At least 4 hours of weekly contact with patient
* Willing to participate in in-person assessments
* -Interested in a family education program for schizophrenia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-03; Primary Completion 2005-12 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Patient BPRS Total Score | baseline, 6 month, 12 month
  Mean total of Brief Psychiatric Rating Scale Score ( BPRS; adapted in Ventura et al, 1993) rated through patient interview. Range is 1-7, with high scores indicating more psychopathology.
Patient Hospitalization | 12 months of study
  Yes/No classification of hospitalization using all sources of data collected in the year

SECONDARY OUTCOMES:
BPRS Psychosis Subscale Score | baseline, 6 month, 12 month
  Mean total of Brief Psychiatric Rating Scale psychosis subscale Score ( BPRS; adapted in Ventura et al, 1993) rated through patient interview. Range is 1-7, with high scores indicating more psychopathology.
Relative Anxiety on the BSI | baseline, 6 months, 12 months
  Relative self-report on the anxiety subscale of the Brief Symptom Inventory (BSI; Derogatis, 1993). Range is 1-5, with high scores indicating more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley M Glynn, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

REFERENCES:
- [Result] Glynn SM, Randolph ET, Garrick T, Lui A. A proof of concept trial of an online psychoeducational program for relatives of both veterans and civilians living with schizophrenia. Psychiatr Rehabil J. 2010 Spring;33(4):278-87. doi: 10.2975/33.4.2010.278.287. PMID 20374986